CLINICAL TRIAL: NCT02378779
Title: Consultations Reason for Genital, Urinary or Psychological Humans in General Practice
Acronym: GETUP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Multiple reminders were carried out but despite these measures, the GP has not enough participated .
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GETUP
Record Dates: First submitted 2015-02-03; First posted 2015-03-04 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Premature Ejaculation
Keywords: Premature ejaculation; general practice; sexual dysfunction
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: This study is a multicenter trial. Patients will be followed either by GPs from the interventional group who trained in communication skills or by the control group who never participated. The distribution of general practitioners in the groups is done thanks random draw .
Masking Description: The study is based on the participation of general practitioners in a training, the test is necessarily open for doctors. However patients will not know if their doctor has received training and will be blinded .
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional GP : GP trainned in communication skills (Other): The subjects have to answer to the questionary SF12 on pre and post consultation to evaluate the quality of life.
  He must so answer to the questionary PEDT. Then the interventional GP group must use one of the six strategies to approach the subject of premature ejaculation.
  There three strategies of attitude (Total attention, Humour, Take the drama out) and three investigative strategies (Question about premature ejaculation, Symptoms of premature ejaculation, Help to verbalize).
  Interventions: Other: Questionary SF12 and PEDT (Premature Ejaculation Diagnostic Tool); Other: Total attention; Other: Humour; Other: Take the drama out; Other: Question about premature ejaculation; Other: Symptoms of premature ejaculation; Other: Help to verbalize
- Usual care : GP did not trainnd in communication skills (Other): The subjects have to answer to the questionary SF12 on pre and post consultation to evaluate the quality of life.
  He must so answer to the questionary PEDT. This classical GP group make a classical consultation like each day without use any strategies to speak about
  Interventions: Other: Questionary SF12 and PEDT (Premature Ejaculation Diagnostic Tool)

INTERVENTIONS:
Other: Questionary SF12 and PEDT (Premature Ejaculation Diagnostic Tool) — The SF-12 was designed to measure general health status from the patient's point of view (12 questions are asking to the patients) and the PEDT questionnaire is a self-assessment questionnaire to diagnose premature ejaculation (5 questions are asking to the patients).
Other: Total attention — Total attention of the GP to approach the subject of premature ejaculation during all the consultation
  Arms: Interventional GP : GP trainned in communication skills
Other: Humour — Use the humour to approach the subject of premature ejaculation
  Arms: Interventional GP : GP trainned in communication skills
Other: Take the drama out — Take the drama out to approach the subject of premature ejaculation
  Arms: Interventional GP : GP trainned in communication skills
Other: Question about premature ejaculation — Question about premature ejaculation during the GP consultation
  Arms: Interventional GP : GP trainned in communication skills
Other: Symptoms of premature ejaculation — GP's observation about signs of premature ejaculation
  Arms: Interventional GP : GP trainned in communication skills
Other: Help to verbalize — Help for the patient to speak about premature ejaculation
  Arms: Interventional GP : GP trainned in communication skills

SUMMARY:
Many male patients complain about their ejaculation: 21-30% of men aged between 18 and 59 have admitted suffering from a decrease in, or loss of control of, their ejaculation. The quality of life of patients and their partners is impaired compared to men not suffering from premature ejaculation. Economically, the impact of the disease are significant. In the year preceding the detection of premature ejaculation patients visit twice their physician. The majority of men interviewed anonymously, in their General Practitioner's ( GP's) waiting room, considered it important to talk with their GP about their sexual concerns. Almost half of them preferred that their GP initiate any discussions about sexuality. More than two thirds of the respondents would have liked their GP to signal his or her open-mindedness by directly addressing sexual topics during the consultation. In 2008 a qualitative study brought to the fore the strategies used by GPs to initiate the discussion on premature ejaculation . GPs who mentioned premature ejaculation with their patient described three attitude-related strategies and three investigative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male patients overbetween 18 and 80 years old and
* Patients consulting for a sexual, urogenital or psychological reason according to Interntational Classification of Primary Care (ICPC-2) will be included.

Exclusion Criteria:

* Patients consulting for Aanother reason for visiting thethan urogenital pattern, sexual or psychological
* Nonunderstanding of the French language
* Patients with psychiatric disorders affecting judgement
* Patient refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
The impact of training general practitioners in communication skills | Day 0 - 4 weeks
  The impact of training general practitioners in communication skills on the rate of patients bringing up the topic of premature ejaculation with their GP. To measure the proportions of patients bringing up the topic of premature ejaculation with their GP, the GPs in the two groups were asked to fill in a questionnaire after the consultation on whether the topics tackled were genital, urinary or psychological. The aim of detailing the different topics broached was to avoid contamination bias in the control group.

SECONDARY OUTCOMES:
Evaluation of quality of life | Day 0 - 4 weeks
  The quality of life will be evaluated with the SF-12 health assessment scale. The SF-12 was designed to measure general health status from the patient's point of view. The SF-12 includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Marie BARAIS, GP, Principal Investigator — GP department, ERCR SPURBO
Locations (23):
- France (23):
  - Cabinet médical, Ambert
  - Cabinet médical - 89 Bis Rue de la Calade, Assas
  - Cabinet médical, Augerolles
  - Cabinet médical, Avermes
  - Cabinet médical - Esplanade Mitterrand 5, Bellerive-sur-Allier
  - Cabinet de médecine générale, Brest
  - Cabinet du 122 rue Paul Masson, Brest
  - Cabinet médical Place J. London, Brest
  - Cabinet médical, Clarensac
  - Cabinet médical, Fleury
  - Pôle universitaire de Lanmeur, Lanmeur
  - Cabinet médical, Le Mayet-de-Montagne
  - Cabinet médical, Le Puy-en-Velay
  - Cabinet médical, Lempdes-sur-Allagnon
  - Cabinet médical du 38 Bd 1848, Narbonne
  - Cabinet de médecine générale, Ondres
  - Cabinet de médecine générale, Pont-de-Buis-lès-Quimerch
  - Cabinet médical du 5 Descente des Oliviers, Restinclières
  - Cabinet médical, Saint-Nicolas-du-Pélem
  - Groupe médical Tourren, Saint-Vincent-de-Tyrosse
  - Cabinet de médecine générale, Saubrigues
  - Cabinet médical, Thézan Les Béziers
  - Cabinet médical - 39 rue Saint Philibert, Trégunc

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After result publication
Access Criteria: The data that will support the findings of this study will be available when the findings will be published in a peerreview journal, from the corresponding author, upon reasonable request

REFERENCES:
- [Derived] Barais M, Vaillant Roussel H, Costa D, Derriennic J, Pereira B, Cadier S. Premature ejaculation in primary care: communication strategies versus usual care for male patients consulting for a sexual, urogenital or psychological reason - GET UP: study protocol for a cluster randomised controlled trial. Trials. 2018 Nov 12;19(1):622. doi: 10.1186/s13063-018-2947-2. PMID 30419940